CLINICAL TRIAL: NCT07208656
Title: The Impact of Medical TV Drama in Improving Literacy on Neurocysticercosis: An Online Open-Label Two-Arm Randomized Controlled Trial
Brief Title: The Impact of Medical TV Drama in Improving Literacy on Neurocysticercosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cephas Health Research Initiative Inc, Ibadan, Nigeria (Network)
Responsible Party: Principal Investigator, Emeka Okeke, Dr., Cephas Health Research Initiative Inc, Ibadan, Nigeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CUL25/NCC/001
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Neurocysticercosis; Health Literacy; Epilepsy
MeSH Terms: conditions — Neurocysticercosis; Epilepsy

STUDY DESIGN:
Intervention Model Description: Two-arm, open-label, randomized controlled trial with parallel assignment.
Masking Description: This is an open-label trial; no blinding was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (House M.D. Episode) (Experimental): Participants in this arm will watch a selected episode of the medical television drama House M.D. (Season 1, Episode 1), which features a dramatized case of neurocysticercosis. The intervention is designed to provide narrative-based exposure to information relevant to the disease. Participants will complete pre- and post-intervention questionnaires assessing knowledge, motivation, and credibility.
  Interventions: Behavioral: Medical TV Drama Episode (House M.D.)
- Control (No Episode) (No Intervention): Participants in this arm will not receive any exposure to medical television content during the study period. They will complete the same pre- and post-intervention questionnaires as the intervention group, allowing comparison of changes in knowledge, motivation, and credibility.

INTERVENTIONS:
Behavioral: Medical TV Drama Episode (House M.D.) — Participants in the experimental group will watch a selected episode of the medical drama House M.D. (Season 1, Episode 1), which includes a dramatized storyline relevant to neurocysticercosis. The episode is intended to deliver narrative-based health education. After viewing, participants will complete post-test questionnaires assessing changes in knowledge, motivation, and credibility compared to pre-test results.
  Other Names: House M.D. Season 1, Episode 1
  Arms: Intervention (House M.D. Episode)

SUMMARY:
This randomized controlled trial evaluates whether exposure to a medical television drama improves knowledge of neurocysticercosis (NCC) among young adults. Sixty participants aged 18-35 will be randomly assigned to either an intervention group, which will watch a medically relevant TV episode (House M.D., Season 1, Episode 1), or a control group with no media exposure. Both groups will complete pre- and post-test questionnaires assessing knowledge of NCC. The primary outcome is change in NCC-related knowledge. Secondary outcomes include motivation to seek further health information and perceived credibility of the media source

DETAILED DESCRIPTION:
Neurocysticercosis (NCC) is a parasitic infection of the central nervous system caused by the larval stage of Taenia solium, the pork tapeworm. It is one of the leading preventable causes of epilepsy worldwide, particularly in low- and middle-income countries (LMICs). Despite this, awareness and understanding of NCC remain low among young adults, who often play a key role in disseminating health information within their families and communities. Conventional health education efforts have had limited success in increasing public literacy about NCC, underscoring the need for innovative, engaging communication strategies.

This study uses an open-label, two-arm randomized controlled trial design to evaluate whether exposure to a medical television drama can improve knowledge of NCC among young adults. The trial will be conducted entirely online to enable participation from a geographically diverse population and to reflect modern media consumption patterns. After providing electronic informed consent, eligible participants will be randomly assigned to either an intervention or control group in a 1:1 ratio using a computer-generated allocation process to ensure randomization integrity.

Participants in the intervention group will watch House M.D., Season 1, Episode 1 - a medically themed television episode featuring a dramatized case of parasitic brain infection with conceptual relevance to NCC. The control group will not view the episode during the study period but will be offered access to the same content after data collection is complete. Both groups will complete structured online questionnaires before and after the intervention period to measure changes in NCC-related knowledge and attitudes. These questionnaires have been developed and validated through expert review and pilot testing.

The trial's primary objective is to determine whether viewing the medical TV drama improves knowledge of NCC, as measured by changes in pre- and post-intervention knowledge scores. Secondary objectives include assessing participants' motivation to learn more about NCC and their perception of the credibility of the TV drama as an educational resource. Statistical analyses will include paired and independent t-tests (or corresponding non-parametric tests where appropriate), with significance set at p < 0.05.

Data will be collected securely using encrypted online survey platforms. All responses will be anonymized, and no personally identifiable information will be stored. Data access will be limited to the research team, and all procedures will comply with international data protection standards.

This trial is designed in accordance with the CONSORT guidelines for randomized behavioral and educational interventions. Ethical approval has been obtained from the Research Ethics Committee of Caleb University, Nigeria, and the study will adhere to the principles outlined in the Declaration of Helsinki (1964). Participation is voluntary, and participants may withdraw at any time before data analysis without consequence.

This research is innovative in its use of entertainment-education as a vehicle for improving disease literacy. By evaluating the effect of a medical TV drama on public knowledge of NCC, the study aims to provide evidence for scalable, cost-effective, and culturally adaptable strategies for health communication in resource-limited settings. The findings are expected to contribute to global public health education efforts, particularly those addressing neglected parasitic diseases and preventable causes of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 35 years
* Proficient in English (reading and comprehension)
* Has access to a stable internet connection
* Possesses a screen-enabled device (e.g., smartphone, tablet, or computer)
* Has access to the Netflix streaming platform

Exclusion Criteria:

* Has formal education in medical or health sciences
* Has a prior diagnosis of neurocysticercosis (NCC)
* Has previously participated in any NCC-related health literacy or awareness program
* Lacks access to the Netflix movie platform
* Below 18 years or above 35 years of age

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in Neurocysticercosis (NCC) Knowledge Score | Baseline and immediately post-intervention (within 1 hour)
  Knowledge of neurocysticercosis (NCC) will be assessed using the Neurocysticercosis Knowledge Questionnaire, a 10-item multiple-choice instrument developed for this study. Each correct answer is scored as 1 point, and each incorrect or "I don't know" response is scored as 0 points. The total score represents the sum of correct answers, with a minimum possible score of 0 and a maximum possible score of 10. Higher scores indicate better knowledge of NCC across domains such as cause, transmission, symptoms, prevention, and treatment. The primary outcome is the change in total knowledge score from baseline (pre-test) to immediately post-intervention, compared between the intervention and control groups

SECONDARY OUTCOMES:
Retention of Neurocysticercosis Knowledge | 4 weeks post-intervention.
  Knowledge retention will be assessed using the Neurocysticercosis Knowledge Questionnaire, the same 10-item multiple-choice instrument used at baseline and immediately post-intervention. Each correct answer is scored as 1 point, and incorrect or "I don't know" responses are scored as 0 points. The total score is the sum of correct responses, with a minimum possible score of 0 and a maximum possible score of 10. Higher scores indicate better retention of NCC knowledge.
  The outcome measure is the change in total knowledge score from baseline (pre-test) to 4 weeks post-intervention, as well as between-group differences in retained knowledge over time.
Perceived Credibility of the Medical TV Drama | Immediately post-intervention (within 1 hour).
  Perceived credibility of the medical TV drama as a health information source will be measured using the Perceived Credibility of Health Media Scale, a 5-item Likert-type scale adapted for this study. Each item is rated from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), assessing dimensions such as trustworthiness, accuracy, and believability of the episode's medical content. Scores for all items will be summed to produce a total credibility score, with a minimum possible score of 5 and a maximum possible score of 25. Higher scores indicate greater perceived credibility and trust in the medical TV drama as a reliable health education resource.
  The outcome measure is the mean total credibility score immediately following the intervention, compared between the intervention and control groups.
Motivation to Seek Further Health Information | Immediately post-intervention (within 1 hour).
  Participants' motivation to seek additional information about neurocysticercosis (NCC) will be assessed using the Motivation to Seek Health Information Scale, a single-item 5-point Likert-type measure adapted for this study. Participants will rate their likelihood of looking for more information about NCC following the intervention, with response options ranging from 1 ("Not at all likely") to 5 ("Extremely likely"). Scores range from 1 to 5, where higher scores indicate greater motivation to seek additional health information.
  The outcome will be reported as the mean motivation score immediately post-intervention and compared between the intervention and control groups.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.